CLINICAL TRIAL: NCT00130403
Title: Open-Label Study to Determine How Prior Therapy With Alendronate or Risedronate in Postmenopausal Women With Osteoporosis Influences the Clinical Effectiveness of Teriparatide
Brief Title: OPTAMISE: Clinical Effectiveness of Teriparatide After Alendronate or Risedronate Therapy in Osteoporotic Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Procter and Gamble (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMR4003B_4034; EudraCT # :2004-002317-37
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Risedronic Acid

INTERVENTIONS:
Drug: risedronate sodium

SUMMARY:
To determine how prior therapy with alendronate or risedronate in postmenopausal women with osteoporosis influences the clinical effectiveness of teriparatide; The primary objective of the study is to compare the teriparatide (human, recombinant PTH[1-34])-associated change from baseline in a marker of bone formation, N-terminal propeptide of type I collagen (P1NP), between subjects previously treated with risedronate and those previously treated with alendronate.

DETAILED DESCRIPTION:
All subjects will be treated with teriparatide (human, recombinant PTH[1-34])(human, recombinant PTH[1-34]), 20 microgram subcutaneously daily for 12 months. Subjects will consist of 290 postmenopausal women previously treated with either risedronate or alendronate for at least 24 months. An approximately equal number of subjects will have been previously treated with risedronate and alendronate, and the subjects will be balanced with regard to duration of previous treatment.

ELIGIBILITY:
ELIGIBILITY CRITERIA include:

* Post-menopausal women who have used risedronate or alendronate continuously for at least 24 mos prior to enrollment
* Dosing regimens allowable are continuous (ie, uninterrupted) daily or weekly formulations of risedronate (5 mg once daily [OD] or 35 or 30 mg once a week [OAW]) or alendronate (10 mg OD or 70 mg OAW), for a minimum of 24 months prior to enrollment into study
* Lumbar spine or total hip BMD T-score 1ess than or equal to -2.0 and >/= 1 prevalent osteoporotic fracture, or lumbar spine or total hip BMD T-score less than or equal to -2.5 with or without and >/= 1 prevalent osteoporotic fracture. The qualifying values must be documented prior to enrollment
* Vitamin D (25-hydroxyvitamin D) between 16 ng/ml and 80 ng/ml
* Urine NTX <50 nmol/mmol creatinine (to assure treatment compliance and bone turnover is in the pre-menopausal range)

EXCLUSION CRITERIA include:

* Impaired renal function, demonstrated by creatinine clearance < 30 ml/min
* Any condition or disease that may interfere with the evaluation of at least 2 lumbar vertebrae (not necessarily contiguous), determined in a screening radiograph by a radiologist at the central facility (eg, confluent aortic calcifications, severe osteoarthritis, spinal fusion, lumbar spine fractures)
* Depot injection vitamin D >10,000 IU in the past 9 months prior to starting the investigational product
* Treatment with antiresorptive agents other than risedronate, alendronate, and hormone replacement therapy within the last 36 months before study entry (ie, ibandronate, pamidronate, etidronate, raloxifene, clodronate, or zoledronate)
* Use of combination alendronate and risedronate, either simultaneously or sequentially, within 60 months prior to enrollment, or use of any anti-resorptive agent in combination with risedronate or alendronate

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2004-03; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Compare the PTH-associated change from baseline at Month 3 of procollagen peptide P1NP, in subjects previously treated with Risedronate or Alendronate | at Month 3

SECONDARY OUTCOMES:
Compare changes from baseline for subjects previously treated with Risedronate or Alendronate for: P1NP & other biomarkers including bone-specific alkaline phosphatase, osteocalcin, serum CTX, urine NTX | at 0.5, 1, 2, 3, 4, 5, 6, & 12 months of treatment
Compare changes from baseline for subjects previously treated with Risedronate or Alendronate for: Lumbar spine & hip BMD measured by DXA | after 6 & 12 months of treatment
Compare changes from baseline for subjects previously treated with Risedronate or Alendronate for: Bone quality parameters captured by central quantitative computed tomography (QCT) | after 12 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Meeves, PharmD, MBA, Study Director — Sanofi
Locations (7):
- sanofi-aventis, US, Bridgewater, New Jersey, United States
- sanofi-aventis, Australia, Cove, New South Wales, Australia
- sanofi-aventis, Belgium, Diegem, Belgium
- sanofi-aventis, Canada, Laval, Quebec, Canada
- sanofi-aventis, France, Paris, France
- sanofi-aventis, Netherlands, Gouda, Netherlands
- sanofi-aventi, UK, Guildford, Surrey, United Kingdom

REFERENCES:
- [Derived] Miller PD, Delmas PD, Lindsay R, Watts NB, Luckey M, Adachi J, Saag K, Greenspan SL, Seeman E, Boonen S, Meeves S, Lang TF, Bilezikian JP; Open-label Study to Determine How Prior Therapy with Alendronate or Risedronate in Postmenopausal Women with Osteoporosis Influences the Clinical Effectiveness of Teriparatide Investigators. Early responsiveness of women with osteoporosis to teriparatide after therapy with alendronate or risedronate. J Clin Endocrinol Metab. 2008 Oct;93(10):3785-93. doi: 10.1210/jc.2008-0353. Epub 2008 Aug 5. PMID 18682511